CLINICAL TRIAL: NCT07288593
Title: Insomnia, Nightmares, and Sympathetic Hyperactivity Intervention in the warfiGHTer (INSIGHT)
Brief Title: INSIGHT: Insomnia, Nightmares, and Sympathetic Hyperactivity Intervention
Acronym: INSIGHT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: University of Minnesota (Other); Walter Reed National Military Medical Center (U.S. Federal Agency); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other); The Geneva Foundation (Other); Applied Physics Laboratory (Unknown); National Intrepid Center of Excellence (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: USUHS.2024-136
Record Dates: First submitted 2025-12-10; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Nightmare; Insomnia; PTSD; TBI; Sleep Disorder (Disorder); REM Behavior Disorder
Keywords: Nightmares; Wearables; Intervention; Sleep quality; Hyperarousal; Insomnia; PTSD; Healthy Participants
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Stress Disorders, Post-Traumatic; Sleep Wake Disorders; REM Sleep Behavior Disorder

STUDY DESIGN:
Intervention Model Description: This study uses a double-blind, randomized, sham-controlled interventional model to test whether the NightWare smartwatch improves sleep quality in warfighters with insomnia and symptoms of sympathetic hyperactivity. Eligible participants from Phase 1 enter a 30-day at-home intervention and are randomly assigned to receive either an active NightWare device or an identical sham device. Neither participants nor study staff know the assignment. All participants wear multiple validated physiological sensors and complete brief daily surveys to measure sleep, autonomic activity, mood, and treatment response. This design allows objective comparison of active versus sham stimulation and supports development of biomarker-based predictors of treatment effectiveness.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Research Coordinators, Research Assistants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control Arm (Sham Comparator): Participants assigned to the sham intervention receive an outwardly identical NightWare smartwatch that does not deliver haptic interventions in response to stress physiology. The sham device collects the same passive physiological data but does not actively attempt to modify sleep or autonomic activity. This arm controls for placebo effects, device expectations, and nightly wear. Participants follow the same 30-day procedures, including daily surveys and physiological sensor wear, ensuring all aspects of participation are identical except for the therapeutic haptic function.
  Interventions: Device: Sham (No Treatment)
- Intervention Arm (Experimental): Participants assigned to the active intervention receive a functioning NightWare smartwatch configured to detect physiological signs of sympathetic activation during sleep, such as heart-rate spikes and movement patterns. When these stress signals exceed a preset threshold, the device delivers brief, gentle haptic vibrations designed to interrupt escalating autonomic arousal without fully awakening the user. The goal is to reduce nighttime sympathetic hyperactivity, improve sleep continuity, and alleviate insomnia symptoms. Participants wear the device nightly for 30 days and complete daily surveys and physiological monitoring to assess treatment effects.
  Interventions: Device: NightWare smartwatch configured to detect physiological signs of sympathetic activation during sleep, such as heart-rate spikes and movement patterns.

INTERVENTIONS:
Device: NightWare smartwatch configured to detect physiological signs of sympathetic activation during sleep, such as heart-rate spikes and movement patterns. — Participants assigned to the active intervention receive a functioning NightWare smartwatch configured to detect physiological signs of sympathetic activation during sleep, such as heart-rate spikes and movement patterns. When these stress signals exceed a preset threshold, the device delivers brief, gentle haptic vibrations designed to interrupt escalating autonomic arousal without fully awakening the user. The goal is to reduce nighttime sympathetic hyperactivity, improve sleep continuity, and alleviate insomnia symptoms. Participants wear the device nightly for 30 days and complete daily surveys and physiological monitoring to assess treatment effects.
  Arms: Intervention Arm
Device: Sham (No Treatment) — NW device that does not deliver any intervention
  Arms: Control Arm

SUMMARY:
The INSIGHT study is a multi-site clinical research program designed to examine how insomnia and symptoms of sympathetic hyperactivity impair sleep, cognition, and physiological restoration in warfighters, and to evaluate whether a wearable therapeutic device can improve these outcomes. Warfighters with a history of traumatic brain injury, post-traumatic stress disorder, or chronic operational stress commonly report disrupted sleep accompanied by manifestations of nocturnal sympathetic activation such as diaphoresis, palpitations, hyperarousal, and nightmares. These symptoms erode sleep quality, reduce cognitive performance, and undermine psychological resilience and operational readiness. Insomnia is two to three times more common in military populations than in civilians, and both TBI and PTSD independently elevate the risk for dysregulated autonomic tone. Excessive sympathetic activity during REM sleep disrupts the normally quiescent locus coeruleus state required for adaptive emotional processing and may contribute to the genesis of nightmares. Excessive sympathetic tone may also interfere with deep NREM-dependent glymphatic clearance, a recently discovered mechanism that supports cognitive restoration and metabolic waste removal. Yet, no study has comprehensively linked these physiological processes in warfighters or evaluated whether wearable-derived autonomic measures can meaningfully stratify insomnia phenotypes. The INSIGHT protocol addresses this gap through a two-phase design integrating multimodal biomarker collection, wearable technology validation, advanced imaging, and a randomized controlled intervention. Phase 1 enrolls 250 participants (50 healthy controls and 200 poor sleepers with or without PTSD and TBI) who undergo structured screening, cognitive testing, and detailed baseline assessments before completing a 2-week at-home data collection period. During this period, participants wear a suite of devices, including EEG headbands, ECG patches, PPG-based sensors, accelerometry rings, blood pressure devices, temperature sensors, and smartwatches, to capture autonomic activity, sleep architecture, cardiovascular and respiratory variability, movement, sudomotor activity, and circadian body temperature patterns. Ecological momentary assessments administered three times daily track fluctuations in sleep quality, mood, PTSD symptoms, and daytime functioning, while urine samples collected on the final three days allow for biochemical analysis of hormonal and sympathetic biomarkers. After the at-home period, all participants complete an overnight in-lab polysomnogram combined with fNIRS to measure sleep stages, autonomic dynamics, cerebral hemodynamics, and glymphatic signatures. A subset of participants also completes an optional overnight MRI with simultaneous EEG following controlled sleep deprivation, enabling state-of-the-art imaging of human glymphatic activity using the MAGNUS MRI platform. This optional visit provides unprecedented insight into how TBI, PTSD, and insomnia alter the physiology of sleep-dependent brain fluid dynamics. In Phase 2, all poor sleepers enter a double-blind, sham-controlled, 30-day randomized trial testing the therapeutic potential of the NightWare smartwatch. NightWare detects sympathetic surges during sleep through heart rate elevations and movement patterns and delivers brief haptic vibrations aimed at interrupting escalating autonomic arousal. Although originally cleared for nightmare treatment, its mechanism is well suited for SNH-related insomnia more broadly. Participants use the device daily while continuing EMA surveys, wearable monitoring, and cognitive assessments, generating rich physiological and behavioral data throughout the intervention. The primary goal is to determine whether reducing nocturnal sympathetic spikes leads to measurable improvements in sleep quality, autonomic stability, daytime functioning, and symptom burden. In parallel, Phase 2 data enable development of the Multi-Organ Autonomic Index of Sleep, an integrated biomarker model that combines neurological, cardiovascular, respiratory, and dermal signals to predict treatment response and classify insomnia subtypes.

The INSIGHT study will produce the most comprehensive dataset to date linking autonomic physiology, glymphatic function, sleep architecture, wearable-derived biomarkers, cognition, and clinical outcomes in warfighters. By identifying physiological signatures of sympathetic hyperarousal and determining whether a non-pharmacological wearable intervention can meaningfully improve sleep, INSIGHT directly supports Department of Defense priorities to enhance readiness, resilience, and long-term neurological health in service members. Wearable tools capable of monitoring and improving sleep outside the laboratory have the potential to transform both clinical care and operational performance, offering scalable and accessible approaches to restoring sleep and optimizing recovery.

DETAILED DESCRIPTION:
Warfighters with mild traumatic brain injury (mTBI) and often comorbid post-traumatic stress disorder (PTSD) are at particularly high risk for disturbed sleep, which undermines performance, psychological health, immune function, and operational readiness. Insomnia is extremely common in these populations, and many report symptoms consistent with nocturnal sympathetic nervous system hyperactivity (SNH), including diaphoresis, hyperarousal, palpitations, tachypnea, and nightmares, which degrade both sleep quality and duration. Insomnia remains one of the most prevalent sleep disorders and is two to three times more common in military and veteran populations than in civilians, with symptoms often lasting decades. Short-term consequences include slowed reaction time, impaired working and visual memory, reduced verbal fluency, and poorer information processing; these changes correlate with hippocampal subregion atrophy in neuroimaging studies. Long-term outcomes include heightened risk of depression, suicidality, cardiovascular disease, cancer, and nearly double the risk of later-life dementia. TBI and PTSD independently impose similar long-term risks, likely compounding insomnia-related impairments. Notably, treating insomnia can improve cognition and even reverse aspects of cortical atrophy in TBI, suggesting that insomnia may be a modifiable mechanism linking these conditions. Military operational exposures increase vulnerability to SNH, offering a plausible explanation for the elevated burden of insomnia in warfighters. Deployment exposure alone has been shown to double insomnia risk, even after accounting for TBI and PTSD. Chronic stress and repeated sleep deprivation, both common in military environments, can produce long-lasting autonomic nervous system (ANS) imbalance and measurable sympathetic excess, including reduced heart rate variability (HRV). Both TBI and PTSD have been independently associated with peripheral and central markers of sympathetic overactivation, including HRV alterations, cardiovascular changes, sweat responses, hormonal patterns, EEG disturbances, and functional MRI findings, with evidence of synergistic effects. SNH relates to insomnia through abnormal HRV, elevated sleeping heart rate and blood pressure, and increased catecholamines and cortisol. Nightmares represent a particularly strong link between stress, PTSD, and SNH. Brain injury affecting the locus coeruleus (LC) is associated with nightmares, and nightmares themselves reflect sympathetic activation. It is therefore plausible that insomnia complaints in warfighters with chronic stress exposure, PTSD, and/or TBI reflect, in part, underlying SNH. Sympathetic tone supports alertness during wakefulness, but excessive activity during sleep is disruptive. The LC drives the fight-or-flight response and activates networks involved in vigilance and threat detection. In healthy sleep, LC activity decreases substantially. Rapid Eye Movement (REM) sleep, critical for emotional processing and dreaming, requires near-silence of the LC, enabling down-regulation of fear circuitry. Excessive LC activation during REM impairs this emotional "resetting" process and likely contributes to nightmare formation. SNH can also produce dream enactment, hyperarousal, startle responses, and peripheral symptoms such as sweating and palpitations. Deep non-REM (NREM) sleep further requires low LC oscillations to allow high-amplitude EEG slow waves, which drive synaptic downscaling, memory consolidation, hormonal rhythms, and cerebrospinal fluid (CSF) flow. These CSF oscillations support glymphatic clearance, the brain's waste-removal system, recently demonstrated in humans via fMRI-EEG studies. Because NREM slow waves support glymphatic activity, and sympathetic activity suppresses these dynamics, warfighters with SNH may experience reduced glymphatic clearance, yet this hypothesis has never been systematically tested in an insomnia population. Insomnia is heterogeneous, and this heterogeneity contributes to inconsistent findings in the literature. Many conditions mimic insomnia or complicate its presentation, including anxiety disorders, circadian misalignment, obstructive sleep apnea (OSA), chronic pain, and reflux. These confounders may explain why some studies fail to replicate associations between insomnia and SNH. Pharmacological targeting of SNH has shown partial success. Prazosin, an alpha-1 adrenergic antagonist, has improved insomnia, nightmares, and cognition in warfighters with PTSD and TBI, though the largest randomized trial in PTSD nightmares did not show benefit, likely in part due to heterogeneous populations and inadequate screening for confounders. Past studies also lacked objective verification of SNH and relied heavily on subjective questionnaires. Gold-standard physiological measures (EEG, fMRI, autonomic monitoring, respiratory signals, and electrodermal activity) are resource-intensive and typically require in-lab recordings, limiting feasibility for large trials. No validated autonomic biomarker currently exists to stratify insomnia patients by SNH burden, highlighting the urgent need for accessible biomarker development. Wearable and "nearable" technologies offer a promising solution. If validated against gold-standard physiological measures, these devices could dramatically expand the ability to capture autonomic and sleep signals in real-world environments. Wearables are comfortable, low-cost, and reduce the artificiality of lab-based sleep measurement. Modern devices measure movement, cardiac and respiratory variability, EEG signals, and electrodermal activity, making them useful for parsing sympathetic and parasympathetic contributions. Sudomotor activity, captured via smartwatches, uniquely reflects pure sympathetic activation. Combined, wearable-derived biomarkers could provide a multidimensional profile of autonomic tone and help stratify patients, monitor treatment effects, and guide intervention development. New approaches to insomnia treatment are needed, particularly for warfighters experiencing SNH. Insomnia is largely defined by self-report, making it difficult to identify mechanistic subtypes. Cognitive Behavioral Therapy for Insomnia (CBTi) remains the gold standard, but access is limited, treatment requires several weeks, and completion rates among warfighters are low. Medications carry notable side effects and are rarely suitable for long-term use. Stellate ganglion block, which reduces peripheral sympathetic output, has shown benefit in PTSD-related hyperarousal and insomnia but is invasive, expensive, and not widely available. A noninvasive, inexpensive, mechanism-targeted option is needed. The NightWare smartwatch represents a promising therapeutic candidate. NightWare is FDA-cleared for treating nightmares; it detects increases in stress physiology via heart rate and movement and delivers brief haptic vibrations to interrupt escalating sympathetic activation. In a prior randomized controlled trial of 75 warfighters with PTSD, poor sleep quality, and frequent nightmares, both sham and active NightWare groups improved, but individuals who wore the device consistently (≥50% of nights) showed significantly greater improvements in sleep quality and nightmare frequency. However, the prior study lacked physiological monitoring to examine how the haptic intervention interacts with sleep stages or autonomic activity. Because NightWare targets sympathetic spikes, it may benefit a broader population of warfighters with insomnia and SNH, even without frequent nightmares. In clinical settings, 20-30% of warfighters endorse nightmares, but many more report other SNH symptoms. This study therefore proposes the first randomized, double-blind, sham-controlled trial to test NightWare in warfighters with insomnia and physiological signs of SNH. A unique feature of the trial is its integration with extensive wearable monitoring and biomarker collection, allowing the device's physiological effects to be characterized in real time. The research will occur in two phases. Phase 1 characterizes baseline sympathetic activity, sleep, cognitive function, self-reported symptoms, and glymphatic markers using a combination of wearable devices, ecological momentary assessments, urine biomarkers, overnight polysomnography, and optional MRI-EEG imaging. Using a diverse array of validated devices allows researchers to capture complementary data streams, such as continuous temperature, high-resolution ECG, EEG, and autonomic signals, necessary for creating a multidimensional profile of sleep and autonomic function. A subset of participants will also complete a sleep-deprivation MRI session using the MAGNUS MRI system to enhance sleep depth during scanning. Sleep deprivation increases sleep pressure, enhances NREM3 slow-wave activity, and can reveal physiological abnormalities not evident during normal baseline sleep, making it ideal for assessing glymphatic dynamics. Phase 2 enrolls poor sleepers into a 30-day randomized, double-blind intervention with either active or sham NightWare devices, alongside daily wearable monitoring and ecological momentary assessments. By integrating high-temporal-resolution physiological signals with behavioral data and treatment exposure, the study aims to identify which autonomic markers predict treatment response and to develop a "Multi-Organ Autonomic Index of Sleep" capable of stratifying insomnia subtypes for future personalized interventions. Wearable data will also quantify the immediate physiological impact of haptic feedback events, enabling iterative improvement of treatment algorithms. The INSIGHT study will generate one of the most comprehensive datasets ever collected on the relationships among autonomic activity, sleep architecture, glymphatic function, trauma exposure, and treatment responsiveness in military populations. The findings will advance efforts to understand the biological mechanisms underlying insomnia in warfighters, identify objective biomarkers for patient stratification, and develop scalable, nonpharmacological treatments that improve readiness and long-term neurological health.

ELIGIBILITY:
Inclusion Criteria:

* Defense Enrollment Eligibility Reporting System (DEERS) Eligible
* Current or former military service member
* Able to read and understand English language without the use of an interpreter
* Habitual bedtime between 9:00 PM and 1:00 AM
* Aged 18-62 (inclusive)
* Able to commit to study procedures

Exclusion Criteria:

* Use of alpha or beta-receptor active medications or prescribed sleep aids in the last 3 months
* Started use of SNRIs or SSRIs in the last 3 months
* Pregnant
* Receiving ongoing and extensive treatment for a new or acute psychiatric disorder within 90 days, other than routine follow-up and care
* Starting concurrent evidence based psychiatric treatment within the past three months
* Diagnosis of a serious medical condition (i.e., late-stage cancer or heart disease)
* Routine night shift work in the past 3 months
* Unstable neurological disease/autonomic disorders/ heart conditions/psych/ sleep or other unstable disorder as determined by the Principal Investigator/Associate
* Investigators determined by clinical interview by Mini international neuropsychiatric interview and medical health questionnaire
* Excessive alcohol use as determined by the AUDIT-C (AUDIT-C > 3)
* Started using any other medication (prescribed or over-the-counter) for the purpose of improving sleep in the last 90 days (e.g., barbiturates, benzodiazepines, melatonin, natural supplements and herbs, antidepressants, antihistamines, etc.)
* Receiving treatment for substance use disorder within 90 days from the start of the study
* Evidence of moderate or severe Obstructive Sleep Apnea (OSA): Determined by the STOP-BANG questionnaire: STOP-BANG greater than 5 Determined by EMR PSG records: moderate or severe OSA [apnea-hypopnea index (AHI)≥15]
* Clinically significant suicidality as assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Currently participating in other research studies for improving sleep
* Currently participating in other research studies for improving PTSD
* Currently in therapy for the primary purpose of improving sleep (e.g., CBT-I)
* Currently undergoing other treatment to improve sleep (e.g., acupuncture)
* History or diagnosis of any of the following sleep disorders: narcolepsy, shift-work disorder or circadian rhythm disorders
* Prone to problems with venipuncture including fainting, hematoma, and infection
* Moderate and high nicotine dependence based on the Fagerstrom Test for Nicotine Dependence (> 4 on the Fagerstrom Test for Nicotine Dependence) High caffeine dependence based on the Caffeine Dependence Questionnaire (> 30 on the Caffeine Dependence Questionnaire)
* Currently experiencing a neurological disorder (e.g., stroke, Parkinson's, MS, etc.)
* Exclusion for optional MRI visit:

Metal in body that is ferromagnetic / incompatible with MRI or other safety issues and indicated by screen Previous adverse reactions to sleep deprivation Illicit drug use as determined by participant self-report Alcohol in system at time of MRI overnight as determined participant self report Nicotine use in the last 3 months

For poor sleep group:

TBI History of epilepsy or suspected seizure disorder.

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
NW efficacy towards sleep quality improvement | 30 days
  Compare Pittsburgh Sleep Quality Index (PSQI) pre- and post-intervention
Autonomic predictors of response to treatment | 30 days
  Predict response to therapy using a model of baseline sympathetic measurements, a "Multi-organ Autonomic Index of Sleep"(MAIS). This model will predict sleep quality using a composite measure of heart rate variability, electrodermal activity, k-complex EEG occurences, estimated locus coruleus activity, and urine noradrenaline.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Walter Reed National Military Medical Center/Uniformed Services University, Bethesda, Maryland
  - University of Minnesota, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davenport ND, Werner JK. A randomized sham-controlled clinical trial of a novel wearable intervention for trauma-related nightmares in military veterans. J Clin Sleep Med. 2023 Feb 1;19(2):361-369. doi: 10.5664/jcsm.10338. PMID 36305584
- [Background] Naegeli C, Zeffiro T, Piccirelli M, Jaillard A, Weilenmann A, Hassanpour K, Schick M, Rufer M, Orr SP, Mueller-Pfeiffer C. Locus Coeruleus Activity Mediates Hyperresponsiveness in Posttraumatic Stress Disorder. Biol Psychiatry. 2018 Feb 1;83(3):254-262. doi: 10.1016/j.biopsych.2017.08.021. Epub 2017 Sep 7. PMID 29100627
- [Background] Sara SJ. The locus coeruleus and noradrenergic modulation of cognition. Nat Rev Neurosci. 2009 Mar;10(3):211-23. doi: 10.1038/nrn2573. Epub 2009 Feb 4. PMID 19190638
- [Background] George SA, Knox D, Curtis AL, Aldridge JW, Valentino RJ, Liberzon I. Altered locus coeruleus-norepinephrine function following single prolonged stress. Eur J Neurosci. 2013 Mar;37(6):901-9. doi: 10.1111/ejn.12095. Epub 2012 Dec 20. PMID 23279008
- [Background] Lampert R, Tuit K, Hong KI, Donovan T, Lee F, Sinha R. Cumulative stress and autonomic dysregulation in a community sample. Stress. 2016 May;19(3):269-79. doi: 10.1080/10253890.2016.1174847. Epub 2016 Apr 25. PMID 27112063
- [Background] Caldwell JA, Knapik JJ, Shing TL, Kardouni JR, Lieberman HR. The association of insomnia and sleep apnea with deployment and combat exposure in the entire population of US army soldiers from 1997 to 2011: a retrospective cohort investigation. Sleep. 2019 Aug 1;42(8):zsz112. doi: 10.1093/sleep/zsz112. PMID 31106808
- [Background] Raikes AC, Dailey NS, Forbeck B, Alkozei A, Killgore WDS. Daily Morning Blue Light Therapy for Post-mTBI Sleep Disruption: Effects on Brain Structure and Function. Front Neurol. 2021 Feb 5;12:625431. doi: 10.3389/fneur.2021.625431. eCollection 2021. PMID 33633674
- [Background] Sivertsen B, Omvik S, Pallesen S, Bjorvatn B, Havik OE, Kvale G, Nielsen GH, Nordhus IH. Cognitive behavioral therapy vs zopiclone for treatment of chronic primary insomnia in older adults: a randomized controlled trial. JAMA. 2006 Jun 28;295(24):2851-8. doi: 10.1001/jama.295.24.2851. PMID 16804151
- [Background] Leng Y, Byers AL, Barnes DE, Peltz CB, Li Y, Yaffe K. Traumatic Brain Injury and Incidence Risk of Sleep Disorders in Nearly 200,000 US Veterans. Neurology. 2021 Mar 30;96(13):e1792-e1799. doi: 10.1212/WNL.0000000000011656. Epub 2021 Mar 3. PMID 33658328
- [Background] Yaffe K, Vittinghoff E, Lindquist K, Barnes D, Covinsky KE, Neylan T, Kluse M, Marmar C. Posttraumatic stress disorder and risk of dementia among US veterans. Arch Gen Psychiatry. 2010 Jun;67(6):608-13. doi: 10.1001/archgenpsychiatry.2010.61. PMID 20530010
- [Background] Chen PL, Lee WJ, Sun WZ, Oyang YJ, Fuh JL. Risk of dementia in patients with insomnia and long-term use of hypnotics: a population-based retrospective cohort study. PLoS One. 2012;7(11):e49113. doi: 10.1371/journal.pone.0049113. Epub 2012 Nov 7. PMID 23145088
- [Background] Yaffe K, Nettiksimmons J, Yesavage J, Byers A. Sleep Quality and Risk of Dementia Among Older Male Veterans. Am J Geriatr Psychiatry. 2015 Jun;23(6):651-4. doi: 10.1016/j.jagp.2015.02.008. Epub 2015 Feb 21. PMID 25794635
- [Background] Sexton CE, Storsve AB, Walhovd KB, Johansen-Berg H, Fjell AM. Poor sleep quality is associated with increased cortical atrophy in community-dwelling adults. Neurology. 2014 Sep 9;83(11):967-73. doi: 10.1212/WNL.0000000000000774. Epub 2014 Sep 3. PMID 25186857
- [Background] von Ruesten A, Weikert C, Fietze I, Boeing H. Association of sleep duration with chronic diseases in the European Prospective Investigation into Cancer and Nutrition (EPIC)-Potsdam study. PLoS One. 2012;7(1):e30972. doi: 10.1371/journal.pone.0030972. Epub 2012 Jan 25. PMID 22295122
- [Background] Cappuccio FP, Miller MA. Sleep and Cardio-Metabolic Disease. Curr Cardiol Rep. 2017 Sep 19;19(11):110. doi: 10.1007/s11886-017-0916-0. PMID 28929340
- [Background] Cappuccio FP, Cooper D, D'Elia L, Strazzullo P, Miller MA. Sleep duration predicts cardiovascular outcomes: a systematic review and meta-analysis of prospective studies. Eur Heart J. 2011 Jun;32(12):1484-92. doi: 10.1093/eurheartj/ehr007. Epub 2011 Feb 7. PMID 21300732
- [Background] Lin HT, Lai CH, Perng HJ, Chung CH, Wang CC, Chen WL, Chien WC. Insomnia as an independent predictor of suicide attempts: a nationwide population-based retrospective cohort study. BMC Psychiatry. 2018 May 2;18(1):117. doi: 10.1186/s12888-018-1702-2. PMID 29716570
- [Background] Tubbs AS, Perlis ML, Basner M, Chakravorty S, Khader W, Fernandez F, Grandner MA. Relationship of Nocturnal Wakefulness to Suicide Risk Across Months and Methods of Suicide. J Clin Psychiatry. 2020 Feb 25;81(2):19m12964. doi: 10.4088/JCP.19m12964. PMID 32097547
- [Background] Joo EY, Kim H, Suh S, Hong SB. Hippocampal substructural vulnerability to sleep disturbance and cognitive impairment in patients with chronic primary insomnia: magnetic resonance imaging morphometry. Sleep. 2014 Jul 1;37(7):1189-98. doi: 10.5665/sleep.3836. PMID 25061247
- [Background] Erickson EA, Stahlman S, McNellis MG. Insomnia and motor vehicle accident-related injuries, active component, U.S. Armed Forces, 2007-2016. MSMR. 2017 Dec;24(12):2-11. PMID 29328680
- [Background] Olaithe M, Ree M, McArdle N, Donaldson S, Pushpanathan M, Eastwood PR, Bucks RS. Cognitive Dysfunction in Insomnia Phenotypes: Further Evidence for Different Disorders. Front Psychiatry. 2021 Jul 19;12:688672. doi: 10.3389/fpsyt.2021.688672. eCollection 2021. PMID 34349682
- [Background] Mysliwiec V, McGraw L, Pierce R, Smith P, Trapp B, Roth BJ. Sleep disorders and associated medical comorbidities in active duty military personnel. Sleep. 2013 Feb 1;36(2):167-74. doi: 10.5665/sleep.2364. PMID 23372263